CLINICAL TRIAL: NCT05881460
Title: Vibrotactile Coordinated Reset: a Non-invasive Treatment for Parkinson's Disease
Brief Title: Vibrotactile Coordinated Reset: a Non-invasive Treatment for Parkinson's Disease 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Synergic Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25412
Record Dates: First submitted 2023-05-19; First posted 2023-05-31 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This study is a double-blinded, crossover trial, where participants are their own control and receive both active stimulation and sham.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active vibrotactile coordinated reset (Active Comparator): Participants will receive active Vibrotactile Coordinated Reset stimulation.
  Interventions: Device: Active vibrotactile coordinated reset
- Sham vibrotactile coordinated reset (Sham Comparator): Participants will receive inactive Vibrotactile Coordinated Reset stimulation.
  Interventions: Device: Sham vibrotactile coordinated reset

INTERVENTIONS:
Device: Active vibrotactile coordinated reset — Vibrotactile Coordinated Reset delivers vibratory stimulation to the fingertips of each hand. A specific pattern of vibration to each fingertip is delivered which theoretically disrupts abnormal synchrony in the brain.
  Other Names: VT Touch glove
  Arms: Active vibrotactile coordinated reset
Device: Sham vibrotactile coordinated reset — Vibrotactile Coordinated Reset delivers vibratory stimulation to the fingertips of each hand. An inactive pattern of vibration to each fingertip is delivered which theoretically will not have the effects of active vCR.
  Other Names: VT Touch glove
  Arms: Sham vibrotactile coordinated reset

SUMMARY:
The purpose of our study is to evaluate Vibrotactile Coordinated Reset stimulation (vCR) and its effects on motor function in people with Parkinson's disease (PD). vCR will be administered with a device called the Vibrotactile (VT) Touch device. vCR can be used in conjunction with medication and is expected to delay the need to increase dopamine medication. It also provides a more flexible alternative to deep brain stimulation (DBS) in that the vCR therapy can be easily stopped or modified to better suit the patients' needs.

DETAILED DESCRIPTION:
This vCR study will include a crossover design, where participants are their own control and receive both active stimulation and sham, aiding in understanding true treatment effects from vCR.

Current treatments for PD include medications, surgical measures, or a combination of both. However, long term use of medications can result in intolerable side effects, especially at higher doses. Although DBS is FDA approved and an established method to manage symptoms of PD, it is an invasive and expensive procedure and may not improve all symptoms of PD. The team at Synergic Medical Technologies, Inc. developed a non-invasive method of applying vibrotactile stimulation delivered through the fingertips that has the potential of theoretically disrupting abnormal synchrony in the brain and thus alleviate severity in motor symptoms in people with PD.

The purpose of this study is to test the use of vibrotactile stimulation on 30 participants with PD and vCRs effects on motor ability using the VT Touch.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 45-85
2. Diagnosis of idiopathic Parkinson's disease from movement disorders neurologist with the United Kingdom Brain Bank criteria of bradykinesia and one or more of the following: rest tremor, rigidity, and balance problems not from visual, vestibular, cerebellar, or proprioceptive conditions
3. Bilateral, moderate-stage impairment, as defined as Hoehn & Yahr Stages II-IV in the on-medication state
4. Able to walk and stand unassisted
5. Participants must be on a stable regimen of PD medication (at least 4 weeks prior to enrollment)
6. Responsive to levodopa (self-reported)
7. Willing to keep exercise and medication regimen as stable as possible for the duration of the study
8. Able to provide informed consent
9. Independently, or with social support, able to use technology and access virtual meeting if needed to troubleshoot technology
10. Participants must speak English and can communicate with staff
11. Patients live close to or in the area of where the clinic is located and are able to travel to the clinic for all screening and assessment appointments.

Exclusion Criteria:

1. Severe depression or suicide ideation (as assessed with Beck Depression Inventory (BDI), BDI <28, and Columbia Suicide Severity Rating scale (SSRS), C-SSRS < 4)

   *BDI score > 28, indicating severe depression that precludes ability to adhere to protocol. Any subject with such a score will be referred to a Primary Care Physician (PCP) or physician for further evaluation and management of depression. Individuals with a BDI score of 17-28 will be excluded if any of the following conditions are met: (1) individual is suicidal, (2) is in need of depression treatment modification currently or (3) depressive symptoms likely to interfere with adherence to study protocol. Any subject with such a score will be referred to a PCP or physician for further evaluation and management of depression.
2. Presence of other neurological or musculoskeletal disorders as determined by the physician during screening.
3. Participation in another drug, device, biologic, or intervention trial concurrently or within the preceding 2-month
4. Physical limitations unrelated to Parkinson's disease
5. Recent change or addition of psychoactive medications for non-parkinsonian treatments
6. Any kind of brain surgery or neurostimulators
7. Pregnancy, breastfeeding, or lack of reliable contraception in women of childbearing age

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in Movement Disorders Society's Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part 3 | baseline, 2 months, 3 months, 5 months
  Difference in MDS-UPDRS Part 3 from baseline to 2 months between active and sham. Range is 0-72 (18 items with 4 being max for each item), higher being worse

SECONDARY OUTCOMES:
Change in gait speed as measured by Ambulatory Parkinson's Disease Monitoring (APDM) Mobility Lab | baseline, 2 months, 3 months, 5 months
  Difference in APDM gait speed from baseline to 2 months between active and sham
Quality of life improvements | baseline, 2 months, 3 months, 5 months
  Quality of life improvements as measured by the Parkinson's disease Quality of Life questionnaire (PDQ-39)
Change in freezing severity index | baseline, 2 months, 3 months, 5 months
  Change in freezing severity index quantified during a turning in place task and other gait spatio-temporal parameters

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Kraakivk, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science Institution, Portland, Oregon, United States